CLINICAL TRIAL: NCT01052961
Title: Initiating Oseltamivir in Adults Hospitalized With Influenza -- a Study on the Impact of Virological Clearance and Clinical Recovery for Higher-dose Treatment Started Within 96 Hours
Brief Title: A Study on Higher-dose Oseltamivir Treatment's Impact on Viral Clearance and Clinical Recovery in Adults Hospitalized With Influenza
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Nelson Lee, Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUHK 7010015, MV22926
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Influenza; Respiratory Tract Infections
Keywords: severe influenza; hospitalized adults; oseltamivir treatment
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections | interventions — Oseltamivir

ARMS (2):
- Non-intervention arm (No Intervention): patients may receive oseltamivir 75 mg bd for 5 days, decided by the managing physicians
- oseltamivir, higher dose (Active Comparator): oseltamivir 150 mg bd for 5 days for patients presented within 96 hours from onset
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir — oseltamivir 150 mg bd for 5 days
  Arms: oseltamivir, higher dose

SUMMARY:
Adult patients hospitalized with influenza have higher viral loads and more severe illnesses. Thus more aggressive treatment approaches (e.g. higher dose oseltamivir) have been suggested to treat patients suffering from severe influenza infection.

The investigators plan to investigate the impact of higher-dose oseltamivir (150 mg b.d.) treatment on viral clearance and clinical recovery in adult patients hospitalized for severe influenza. Such information may lead to optimization of the management strategy used for these patients.

DETAILED DESCRIPTION:
* The investigators plan to study the impact of higher-dose oseltamivir (150 mg b.d.) treatment on rate of viral load decline and RNA negativity (in nasal and throat swabs, assessed by quantitative RT-PCR assay) and time to clinical recovery in adult patients hospitalized for severe influenza.
* Patients who received intervention (oseltamivir 150 mg b.d. for 5 days) will be compared to those in the non-intervention arm (patients may receive oseltamivir treatment at 75 mg b.d. for 5 days, decided by their managing physicians) in the two respective study sites. Viral load changes and viral clearance will be compared. Clinical progress and time to symptom recovery will be reported. The protocol will be crossed-over to the other site at a defined time frame.
* oseltamivir 150 mg b.d. has been shown to be safe and well-tolerated in earlier clinical trials
* higher-dose treatment has been suggested by health authorities (e.g. WHO) to treat severe influenza infection/pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* confirmed influenza A (H1N1, H3N2) or B infection by IFA or RT-PCR, with a compatible clinical illness
* presented within 96 hours from symptom onset
* age >/= 18 years

Exclusion Criteria:

* lack of consent
* suspected avian influenza
* patients who have received antivirals against influenza prior to admission
* suspected or confirmed oseltamivir resistance
* pre-existing renal impairment, with creatinine clearance <40 ml/min
* pre-existing hepatic failure
* participation in a clinical study involving experimental medication in the past 4 weeks
* pregnant women, or who are attempting to become pregnant, or who are breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
rate of influenza virus load decline and viral RNA negativity upon receiving 5 days of study treatment | during and upon completion of the 5-day study treatment

SECONDARY OUTCOMES:
time to clinical recovery (including symptoms, vital signs, hospital discharge) | during and upon completion of the 5-day study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nelson LS Lee, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Prince of Wales Hospital and Alice Ho Miu Ling Nethersole Hospital, Hong Kong, Hksar, Hong Kong

REFERENCES:
- [Background] Lee N, Chan PK, Hui DS, Rainer TH, Wong E, Choi KW, Lui GC, Wong BC, Wong RY, Lam WY, Chu IM, Lai RW, Cockram CS, Sung JJ. Viral loads and duration of viral shedding in adult patients hospitalized with influenza. J Infect Dis. 2009 Aug 15;200(4):492-500. doi: 10.1086/600383. PMID 19591575
- [Background] Lee N, Cockram CS, Chan PK, Hui DS, Choi KW, Sung JJ. Antiviral treatment for patients hospitalized with severe influenza infection may affect clinical outcomes. Clin Infect Dis. 2008 Apr 15;46(8):1323-4. doi: 10.1086/533477. No abstract available. PMID 18444878
- [Background] Lee N, Wong CK, Chan PK, Lun SW, Lui G, Wong B, Hui DS, Lam CW, Cockram CS, Choi KW, Yeung AC, Tang JW, Sung JJ. Hypercytokinemia and hyperactivation of phospho-p38 mitogen-activated protein kinase in severe human influenza A virus infection. Clin Infect Dis. 2007 Sep 15;45(6):723-31. doi: 10.1086/520981. Epub 2007 Aug 8. PMID 17712756
- [Background] Lee N, Chan PK, Choi KW, Lui G, Wong B, Cockram CS, Hui DS, Lai R, Tang JW, Sung JJ. Factors associated with early hospital discharge of adult influenza patients. Antivir Ther. 2007;12(4):501-8. PMID 17668558
- [Background] Treanor JJ, Hayden FG, Vrooman PS, Barbarash R, Bettis R, Riff D, Singh S, Kinnersley N, Ward P, Mills RG. Efficacy and safety of the oral neuraminidase inhibitor oseltamivir in treating acute influenza: a randomized controlled trial. US Oral Neuraminidase Study Group. JAMA. 2000 Feb 23;283(8):1016-24. doi: 10.1001/jama.283.8.1016. PMID 10697061
- [Background] Nicholson KG, Aoki FY, Osterhaus AD, Trottier S, Carewicz O, Mercier CH, Rode A, Kinnersley N, Ward P. Efficacy and safety of oseltamivir in treatment of acute influenza: a randomised controlled trial. Neuraminidase Inhibitor Flu Treatment Investigator Group. Lancet. 2000 May 27;355(9218):1845-50. doi: 10.1016/s0140-6736(00)02288-1. PMID 10866439
- [Background] World Health Organization. Clinical management of human infection with pandemic (H1N1) 2009: revised guidance. Available at: http://www.who.int/csr/resources/publications/swineflu/clinical_management_h1n1.pdf. Last accessed on 1st Dec, 2009
- [Derived] Lee N, Hui DS, Zuo Z, Ngai KL, Lui GC, Wo SK, Tam WW, Chan MC, Wong BC, Wong RY, Choi KW, Sin WW, Lee EL, Tomlinson B, Hayden FG, Chan PK. A prospective intervention study on higher-dose oseltamivir treatment in adults hospitalized with influenza a and B infections. Clin Infect Dis. 2013 Dec;57(11):1511-9. doi: 10.1093/cid/cit597. Epub 2013 Sep 17. PMID 24046309